CLINICAL TRIAL: NCT06597903
Title: A Pilot Monocentric, Open Phase II Study to Investigate the Efficacy and Safety of a New Gut Cleansing Solution ("Low Dose Bowel Prep") in 30 Patients Submitted to Colonoscopy
Brief Title: A Monocentric Study to Investigate a New Low Dose Oral Gut Cleansing Solution
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NRL994-01/2000
Record Dates: First submitted 2015-06-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — MoviPrep

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (1):
- NRL994 low dose bowel prep (LDBP) (Experimental): Patients given two doses of NRL994, one on the evening before and one on the morning of their scheduled colonoscopy. Degree of gut cleansing was rated by the colonoscopist and an independent reviewer. Volume of fluid aspirated during colonoscopy and weight of stools/volume of urine from start of cleansing to start of colonoscopy were also measured. Number of patients who reached clear effluent evaluated.
  Interventions: Drug: NRL994

INTERVENTIONS:
Drug: NRL994 — In the afternoon/evening before colonoscopy: 1 litre solution plus 0.5 litre clear fluid.
  Day of colonoscopy: 1 litre solution plus at least up to 1 litre clear liquid.
  Other Names: Low dose bowel prep (LDBP); MOVIPREP

SUMMARY:
A first study at one centre, with a new oral gut cleansing solution, NRL994, in patients who were going to have a colonoscopy. The study was to find out how well the new "Low Dose Bowel Prep" (LDBP) worked, and whether it was safe to use.

DETAILED DESCRIPTION:
A pilot monocentric, open phase I study to investigate the efficacy and safety of a new oral gut cleansing solution NRL994 in patients submitted to colonoscopy.

The study was carried out as an open, uncontrolled investigation in a group of 36 in-patients scheduled for colonoscopy. Patients were enrolled one or two days prior to the endoscopic procedure. Gut cleansing started in the evening prior to the intervention when the first dose of LDBP was taken; bowel preparation was continued in the morning of the day of colonoscopy when the second dose was taken. A patient's participation in the study ended after completion of the endoscopic procedure.

A dose of NRL994 was diluted in 1000 mL of water and consisted of 100 g PEG 3350, 7.5 g sodium sulphate, 4.7 g ascorbic acid, 5.9 g sodium ascorbate, 46 mmol sodium chloride, and 12.46 mmol potassium chloride. The product was flavoured with lemon flavour (2.015 g), anhydrous citric acid (1.565 g), and potassium acesulfame (0.35 g).

Each dose of one litre had to be swallowed within one hour, followed by 500 mL of additional clear fluid.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained prior to inclusion
* Male or female
* Inpatients 18 to 60 years old with indication for complete colonoscopy
* Willing and able to complete the entire procedure and to comply with study instructions
* Females of childbearing potential must employ an adequate method of contraception.

Exclusion Criteria:

* Ileus
* Intestinal obstruction or perforation.
* Toxic megacolon.
* History of any colonic surgery.
* Cardiac Insufficiency (NYHA grad III and IV).
* Ischemic cardio vascular disease.
* Renal insufficiency (creatinine above 1.4 mg/100 ml).
* Cirrhosis of liver (child B or C).
* Known hypersensitivity to polyethylene glycols and/or Vitamin C.
* Concurrent participation in an investigational drug study or participation within 30 days of study entry.
* Females who are pregnant, nursing or planning a pregnancy. Females of child bearing potential not using reliable methods of contraception.
* Subject has a condition or is in a situation which in the investigators opinion may put the subject at significant risk, may confound the study results, or may interfere significantly.
* Abnormal laboratory values (clinically significant) for sodium, potassium, chloride, creatinine and hematocrit
* Untreated or uncontrolled arterial hypertension (max. > 170 mmHg and min > 100 mmgH).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2001-05; Primary Completion 2002-03 (Actual); Study Completion 2002-03 (Actual)

PRIMARY OUTCOMES:
Degree of gut cleansing | Day 0 during colonoscopy
  Degree of gut cleansing in each of five predefined gut segments (rectum, sigmoid colon, descending colon, transverse colon, ascending colon) rated on a 5-level verbal rating scale (VRS) ranging from 4 (very good) to 0 (very bad) by
  1. the physician performing the endoscopic procedure and
  2. by an independent reviewer on the basis of video tapes registered during colonoscopy.
Overall quality of colonic cleansing | Day 0 during colonoscopy
  Overall quality of colonic cleansing as rated on a 3-level VRS with ranks:
  A = very good or good colon cleansing in all five gut segments, B = at least one colon segment with moderate or bad cleansing result, C = very bad cleansing result in at least one colon segment.
Physicians overall judgement of colon preparation | Day 0 during colonoscopy
  Physicians overall judgement of colon preparation as assessed on a 5-level VRS ranging from very good to very bad.
Volume of fluid aspirated (ml) | Day 0 during colonoscopy
  Volume of fluid aspirated from intestinal lumen during colonoscopy.
Stool and urine weight (g) | Day -1 and Day 0 prior to colonoscopy.
  Weight of stools and urine sampled from the beginning of gut preparation until the start of the endoscopic procedure.
Clear effluent | Day -1 and Day 0 prior to colonoscopy.
  Number of patients in whom a clear effluent (containing no residual faecal material) was obtained.
Patient satisfaction - convenience | Day -1 and Day 0 prior to colonoscopy
  Patients overall judgement of convenience of use of LDBP as assessed in the CRF on a on a 5-level VRS ranging from 4 (very good) to 0 (very bad).
Patient satisfaction - taste | Day -1 and Day 0 prior to colonoscopy
  Patients overall judgement of the taste of LDBP as assessed in the CRF on a on a VAS ranging from 0 (very bad) to 100 mm (very good).

SECONDARY OUTCOMES:
Adverse events | Day -1 and Day 0 prior to colonoscopy
  • Occurrence of adverse events;
Global tolerance | Day -1 and Day 0 prior to colonoscopy
  Physicians global assessment of tolerability of LDBP as rated on a 4-level VRS ranging from (excellent) to (bad).
Hematology | Day -2 to Day 0 prior to colonoscopy
  A blood sample was obtained for hematology (hematocrit, hemoglobin, red and white blood cell count, platelet count) at baseline and after intake of the second dose of LDBP just before colonoscopy.
Serum chemistry | Day -2 to Day 0 prior to colonoscopy
  A blood sample was obtained for serum chemistry (electrolytes [sodium, potassium, chloride, bicarbonate], liver enzymes [ASAT, ALAT], total protein, blood urea nitrogen [BUN], creatinine, Quick time) at baseline and after intake of the second dose of LDBP just before colonoscopy.
Urine electrolytes | Day -1 to Day 0 prior to colonoscopy
  Amount of electrolytes (sodium, potassium, calcium) excreted in urine sampled from the beginning of gut preparation until the start of the endoscopic procedure.
Blood pressure (mmHg) | Day -2 to Day 0 after colonoscopy
  Blood pressure was measured at baseline, upon completion of LDBP intake, and after the end of colonoscopy.
Pulse rate (bpm) | Day -2 to Day 0 after colonoscopy
  Pulse rate in beats per minute (bpm) was measured at baseline, upon completion of LDBP intake, and after the end of colonoscopy.
Body weight (kg) | Day -1 prior to LDBP and Day 0 prior to colonoscopy.
  Actual body weight in kilograms (kg) was measured before and after the administration of LDBP.

OTHER OUTCOMES:
Easiness | Day -1 and Day 0 prior to colonoscopy
  Patients overall judgement of convenience of use (easiness) of LDBP as assessed in the diary card on a on a 5-level VRS ranging from 4 (very good) to 0 (very bad).
Palatability | Day -1 and Day 0 prior to colonoscopy
  Patient satisfaction with the palatability (taste and convenience) of the first and the second liter of LDBP cleansing solution ingested as assessed in the diary card on a 5-level VRS ranging from 4 (very good) to 0 (very bad)
  Time Frame:

CONTACTS AND LOCATIONS:
Overall Officials: K-J Goerg, PD Dr. med., Principal Investigator — Dept. of Internal Medicine II, St. Antonius Hospital, Hardt 46, D-42 107 Wuppertal, Germany
Locations (1):
- Med. Klinik der, Wuppertal, Germany